CLINICAL TRIAL: NCT02180295
Title: A Phase III, Double-Blind, Lot-To-Lot Consistency Clinical Trial to Evaluate the Safety, Tolerability and Immunogenicity of V212 in Healthy Adults
Brief Title: A Lot-to-Lot Consistency Study to Evaluate Safety, Tolerability, and Immunogenicity of Inactivated Varicella Zoster Virus (VZV) Vaccine in Healthy Adults (V212-014)
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: V212-014; 2014-001030-29 (EudraCT Number)
Record Dates: First submitted 2014-07-01; First posted 2014-07-02 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Herpes Zoster
MeSH Terms: conditions — Herpes Zoster

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- V212 Lot 1 (Experimental): Approximately 7.5 Units/0.5 mL subcutaneous injection administered in a 4-dose regimen given approximately 30 days apart
  Interventions: Biological: V212 Lot 1
- V212 Lot 2 (Experimental): Approximately 7.5 Units/0.5 mL subcutaneous injection administered in a 4-dose regimen given approximately 30 days apart
  Interventions: Biological: V212 Lot 2
- V212 Lot 3 (Experimental): Approximately 7.5 Units/0.5 mL subcutaneous injection administered in a 4-dose regimen given approximately 30 days apart
  Interventions: Biological: V212 Lot 3

INTERVENTIONS:
Biological: V212 Lot 1 — Inactivated Varicella Zoster Virus vaccine
  Arms: V212 Lot 1
Biological: V212 Lot 2 — Inactivated Varicella Zoster Virus vaccine
  Arms: V212 Lot 2
Biological: V212 Lot 3 — Inactivated Varicella Zoster Virus vaccine
  Arms: V212 Lot 3

SUMMARY:
The study will evaluate the consistency of 3 lots of inactivated VZV vaccine for safety, tolerability, and immunogenicity in healthy adults. The primary hypothesis of the study is that the 3 lots of inactivated vaccine will demonstrate similar immunogenicity at 28 days after the fourth dose.

ELIGIBILITY:
Inclusion Criteria:

* Afebrile (<=100.4 °F [<=38.0 °C]) oral or equivalent on Day 1 before the first vaccination
* Any underlying chronic illness that is not in stable condition
* History of varicella, antibodies to VZV, or residence (for >=30 years) in a country with endemic VZV infection
* Female participants of childbearing potential must have a negative pregnancy test. A female not of reproductive potential has reached natural menopause, or is 6-weeks postsurgical bilateral oophorectomy and/or hysterectomy or bilateral tubal ligation
* Male, or female of childbearing potential who agrees to remain abstinent or use 2 acceptable methods of birth control from 2 weeks before enrollment to 6 months after the last study vaccination

Exclusion Criteria:

* History of allergic reaction to any vaccine component, or an anaphylactic/anaphylactoid reaction to neomycin (not including contact dermatitis to neomycin)
* Prior history of herpes zoster
* History of receipt or expects to receive any varicella or zoster vaccine during the study period
* Is pregnant or breastfeeding, or expects to conceive from 2 weeks before enrollment to 6 months after the last study vaccination
* Has received a live virus vaccine or is scheduled to receive any live virus vaccine from 4 weeks before the first dose of study vaccination and throughout the study
* Has received any inactivated vaccine or is scheduled to receive any inactivated vaccine from 7 days before to 7 days after any study vaccination
* Received immunoglobulin or any blood products or is scheduled to receive them from 5 months before the first dose of study vaccination and throughout the study
* Has participated in an investigational drug or vaccine study within 30 days before enrollment
* Has any acute illness or significant underlying illness that may interfere with interpretation of the study
* Receiving immunosuppressive therapy (including systemic corticosteroid doses exceeding physiological replacement doses within 14 days prior to the first vaccination), except topical, ophthalmic, or inhaled corticosteroids or intra-articular or soft-tissue injections of steroids
* Has known or suspected immune dysfunction

Ages: 50 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2014-07; Primary Completion 2015-03 (Estimated); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
Geometric Mean Titer of VZV Glycoprotein Enzyme-Linked Immunosorbent Assay (gpELISA) Antibody Titers | 28 days postdose 4

SECONDARY OUTCOMES:
Percentage of Participants with a Serious Adverse Experience | Up to 28 days postdose 4

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Derived] de Oliveira Gomes J, Gagliardi AM, Andriolo BN, Torloni MR, Andriolo RB, Puga MEDS, Canteiro Cruz E. Vaccines for preventing herpes zoster in older adults. Cochrane Database Syst Rev. 2023 Oct 2;10(10):CD008858. doi: 10.1002/14651858.CD008858.pub5. PMID 37781954